CLINICAL TRIAL: NCT00579241
Title: Detection of Ultrasound Contrast Signals in the Cerebral Circulation During Stress Echocardiography
Brief Title: Detection of Ultrasound Contrast Signals in the Cerebral Circulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0113-06-FB
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Brain Vascular Disorders; Coronary Artery Disease
MeSH Terms: conditions — Cerebrovascular Disorders; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 Transcranial imaging using Doppler Ultrasound (Experimental): Transcranial imaging using Doppler ultrasound
  Interventions: Procedure: Ultrasound on Temporal Bone

INTERVENTIONS:
Procedure: Ultrasound on Temporal Bone — All Patients undergoing dobutamine stress echocardiography have an intravenous line placed and a continuous infusion of a commercially available contrast agent administered. Prior to contrast infusion, baseline transcranial ultrasound images at 0.4 mechanical index using low mechanical index pulses and color Doppler will be performed and recorded. After this the contrast infusion will begin, and resting cardiac images will occur.

SUMMARY:
To Determine whether transcranial ultrasound can detect the presence of intravenously injected microbubbles used routinely for dobutamine stress echocardiography.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the intravenous microbubbles used to improve border delineation during dobutamine stress echocardiographies (DSE) can be detected within the cerebral circulation.

ELIGIBILITY:
Inclusion Criteria:

* male or female age >19 years of age
* scheduled for a stress echocardiogram
* negative urine pregnancy test within two hours of ultrasound contrast administration required for females of childbearing age unless post-menopausal or with evidence of surgical sterilization
* be conscious and coherent, and able to communicate effectively with trial personnel

Exclusion Criteria:

* pregnant or lactation
* life expectancy of less than 2 months or terminally ill
* Known or suspected hypersensitivity to ultrasound contrast agent used for the study
* complicated hemodynamic instability
* Known left main disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04-27 (Actual); Primary Completion 2009-12-12 (Actual); Study Completion 2009-12-12 (Actual)

PRIMARY OUTCOMES:
Detect abnormalities in cerebral blood flow | immediate
  All Patients undergoing dobutamine stress echocardiography have an intravenous line placed and a continuous infusion of a commercially available contrast agent administered. Prior to contrast infusion, baseline transcranial ultrasound images at 0.4 mechanical index using low mechanical index pulses and color Doppler will be performed and recorded. After this the contrast infusion will begin, and resting cardiac images will occur.

SECONDARY OUTCOMES:
if cerebral vascular disease is detected it would lead to further testing that may better identify abnormalities. | within 30 minutes
  All Patients undergoing dobutamine stress echocardiography have an intravenous line placed and a continuous infusion of a commercially available contrast agent administered. Prior to contrast infusion, baseline transcranial ultrasound images at 0.4 mechanical index using low mechanical index pulses and color Doppler will be performed and recorded. After this the contrast infusion will begin, and resting cardiac images will occur.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska Medicial Center